CLINICAL TRIAL: NCT05376878
Title: Pilot Study to Evaluate 64Cu-DOTA-Trastuzumab Imaging in Patients With HER2+ Breast Cancer With Brain Metastatsis Treated With Fam-Trastuzumab Deruxtecan
Brief Title: An Investigational Scan (64Cu-DOTA-Trastuzumab PET/MRI) in Imaging Patients With HER2+ Breast Cancer With Brain Metastasis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21050; NCI-2022-03220 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21050 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2022-05-03; First posted 2022-05-17 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Breast Carcinoma; Metastatic Malignant Neoplasm in the Brain
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — 64Cu-DOTA-trastuzumab; Magnetic Resonance Spectroscopy; Positron-Emission Tomography; Trastuzumab; PF-05280014; Ogivri; Ontruzant; trastuzumab biosimilar HLX02; trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Treatment ( 64Cu-DOTA-trastuzumab PET/MRI) (Experimental): Patients receive trastuzumab IV over 15 minutes on day 0. Patients then receive 64Cu-DOTA-trastuzumab IV and then undergo PET/MRI scan on day 1. Patients undergo repeat brain MRI every 6 weeks for 24 weeks and then every 9 weeks until disease progression. Patients then receive trastuzumab deruxtecan IV every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Copper Cu 64-DOTA-Trastuzumab; Procedure: Magnetic Resonance Imaging; Device: Positron Emission Tomography; Biological: Trastuzumab; Biological: Trastuzumab Deruxtecan

INTERVENTIONS:
Other: Copper Cu 64-DOTA-Trastuzumab — Given IV
  Other Names: 64Cu-DOTA-Trastuzumab
Procedure: Magnetic Resonance Imaging — Undergo PET/MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Device: Positron Emission Tomography — Undergo PET/MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Biological: Trastuzumab — Given IV
  Other Names: ABP 980; ALT02; Anti-c-ERB-2; Anti-c-erbB2 Monoclonal Antibody; Anti-ERB-2; Anti-erbB-2; Anti-erbB2 Monoclonal Antibody; Anti-HER2/c-erbB2 Monoclonal Antibody; Anti-p185-HER2; c-erb-2 Monoclonal Antibody; HER2 Monoclonal Antibody; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; Herzuma; Kanjinti; MoAb HER2; Monoclonal Antibody c-erb-2; Monoclonal Antibody HER2; Ogivri; Ontruzant; PF-05280014; rhuMAb HER2; RO0452317; SB3; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar ALT02; trastuzumab biosimilar EG12014; Trastuzumab Biosimilar HLX02; Trastuzumab Biosimilar PF-05280014; Trastuzumab Biosimilar SB3; Trastuzumab Biosimilar SIBP-01; Trastuzumab-anns; Trastuzumab-dkst; Trastuzumab-dttb; Trastuzumab-pkrb; Trastuzumab-qyyp; Trazimera
Biological: Trastuzumab Deruxtecan — Given IV
  Other Names: DS-8201; DS-8201a; Enhertu; Fam-trastuzumab Deruxtecan-nxki; WHO 10516

SUMMARY:
This clinical trial examines an investigational scan (64Cu-DOTA-trastuzumab positron emission tomography [PET]/magnetic resonance imaging [MRI]) in imaging patients with HER2+ breast cancer that has spread to the brain (brain metastasis). Diagnostic procedures, such as 64Cu-DOTA-trastuzumab PET/MRI, may help find HER2+ breast cancer that has spread to the brain and determine whether cancer in the brain takes up trastuzumab, which may predict for response to trastuzumab deruxtecan (the standard of care chemotherapy).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the feasibility of 64Cu-DOTA-trastuzumab PET imaging in patients with HER2+ breast cancer metastatic to the brain.

II. Evaluate if HER2+ breast cancer patients with brain metastasis who are responders to fam-trastuzumab deruxtecan have higher maximum standardized uptake value (SUVmax) (minimum over all lesions in the brain) than non-responders.

SECONDARY OBJECTIVE:

I. Evaluate if the minimum SUVmax of all quantifiable lesions in a given patient is associated with time to progression in the brain.

OUTLINE:

Patients receive trastuzumab intravenously (IV) over 15 minutes on day 0. Patients then receive 64Cu-DOTA-trastuzumab IV and then undergo PET/MRI scan on day 1. Patients undergo repeat brain MRI every 6 weeks for 24 weeks and then every 9 weeks until disease progression. Patients then receive trastuzumab deruxtecan IV every 21 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Women with documented metastatic HER2 positive breast cancer (American Society of Clinical Oncology [ASCO] College of American Pathologist [CAP] guidelines) who have brain metastases
* Age > 18 years
* Eastern Cooperative Oncology Group (ECOG) 0-2
* Patients with leptomeningeal disease will be considered eligible
* Planned therapy with fam-trastuzumab deruxtecan
* Left ventricular ejection fraction (LVEF) > 50%
* Absolute neutrophil count (ANC) > 1.5 x 10^9/L
* Platelets > 100 x 10^9/L
* Hemoglobin > 9 g/dL
* Total (T.) bilirubin < 3 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 5 x ULN
* Creatinine clearance > 30 ml/min (by Cockcroft-Gault formula)
* Activated partial thromboplastin time (aPTT) < 1.5 x ULN
* Prior therapy for central nervous system (CNS) disease is allowed, but at least 1 lesion > 1.5 cm is evident on MRI

Exclusion Criteria:

* Need for immediate local intervention for brain metastases
* Noninfectious interstitial lung disease or pneumonitis requiring glucocorticoids
* Clinically significant corneal disease
* Myocardial infarction < 6 months before, congestive heart failure (CHF), unstable angina, or serious cardiac arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Percent of patients with quantifiable 64Cu-DOTA-trastuzumab PET uptake | Until disease progression or death, up to 5 years.
  Percentage of patient with quantifiable 64Cu-DOTA-trastuzumab PET imaging (maximum standardized uptake value[SUVmax]) uptake in brain lesions.
Comparison of average min SUVmax values in responders versus non-responders. | Until disease progression or death, up to 5 years.
  Comparison evaluated using a non-parametric test. The lowest SUVmax (minimum SUVmax) across the lesions will be the primary metric used. Response assessment for CNS disease is determined by MRI of the brain using Response Assessment in Neuro-Oncology (RANO) criteria.

SECONDARY OUTCOMES:
Progression-free Survival | From start of treatment until progression or death from any cause, up to 5 years.
  Estimated using the product-limit method of Kaplan and Meier. Progression defined by any of the following: > 25% increase in sum of the products of perpendicular diameters of enhancing lesions; any new lesion; or clinical deterioration.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne E Mortimer, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States